CLINICAL TRIAL: NCT01808950
Title: Bi-center, Open Label, Non-comparative Trial Exploring Efficacy and Safety of Topical Resiquimod Gel (0.06%) in Patients With Nodular Basal Cell Carcinoma (nBCC)
Brief Title: Efficacy and Safety Trial of Topical Resiquimod Gel (0.06%) in Patients With Nodular Basal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: safety issues
Sponsor: Spirig Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SP848-nBCC-1104
Record Dates: First submitted 2013-03-05; First posted 2013-03-11 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Nodular Basal Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.06% Resiquimod Gel - A (Experimental): * 60 mg gel
  * Once daily prior to normal sleeping hours
  * 5x within 1 week (Monday to Friday) for 4 weeks (at maximum) or until clinical manifestation of skin erosion/crust formation
  Interventions: Drug: 0.06% Resiquimod Gel - A
- 0.06% Resiquimod Gel - B (Experimental): * 100 mg gel
  * Once daily prior to normal sleeping hours
  * 5x within 1 week (Monday to Friday) for 4 weeks (at maximum) or until clinical manifestation of skin erosion/crust formation
  Interventions: Drug: 0.06% Resiquimod Gel - B
- 0.06% Resiquimod Gel - C (Experimental): * 100 mg gel
  * Once daily prior to normal sleeping hours
  * 5x within 1 week (Monday to Friday) for 4 weeks (at maximum) or until clinical manifestation of skin erosion/crust formation
  * The BCC will be pretreated. A shave biopsy (curettage or scraping off the tissue in a broad, superficial, tangential way) will be performed
  Interventions: Drug: 0.06% Resiquimod Gel - C

INTERVENTIONS:
Drug: 0.06% Resiquimod Gel - A — single 60mg dose
  Other Names: CD11301
  Arms: 0.06% Resiquimod Gel - A
Drug: 0.06% Resiquimod Gel - B — single 100mg dose
  Other Names: CD11301
  Arms: 0.06% Resiquimod Gel - B
Drug: 0.06% Resiquimod Gel - C — shave biopsy of BCC followed by single 100mg dose
  Other Names: CD11301
  Arms: 0.06% Resiquimod Gel - C

SUMMARY:
The primary objective is the observation and description of the preliminary efficacy of resiquimod gel 0.06% on a single nodular basal cell carcinoma (nBCC) in a small group of patients.

DETAILED DESCRIPTION:
efficacy assessments:

* Histopathological findings based on the biopsies of the primary tumor location and the tissue excision at the end of trial (histological cure).
* Description of the clinical-therapeutic effect of resiquimod on nBCC (nodular-basal cell carcinoma) by visual inspection (clinical evaluation of treatment area and assessment of complete clinical clearance)
* RNA-analysis (analysis of gene expressions for cytokines, cytotoxic and apoptotic signals)
* Investigator's global judgment of efficacy by means of a 7-point scale

Safety assessments:

* Evaluation of Adverse Events (AEs) and Serious Adverse Events (SAEs)
* Evaluation of local tolerability (local skin reactions as erythema, edema, erosion/ulceration, exsudate, dryness, encrustation) by means of symptom scoring scales (0 = absent, 1 = slight, 2 = moderate, 3 = severe, 4 = very severe).
* Evaluation of systemic tolerability [hematology (erythrocytes, leucocytes including neutrophils, hemoglobin, hematocrit, thrombocytes), blood chemistry (alkaline phosphatase, bilirubin, aspartate transaminase (ASAT), alanine transaminase (ALAT), serum creatinine), vital signs]. The thresholds concerning laboratory abnormalities that determine patient's discontinuation from trial were predefined upfront.
* Evaluation of the number of patients withdrawn from the trial
* Investigator's global judgment of tolerability by means of a 6-point scale
* Photographic documentation of the treatment area

Exploratory parameter:

* C-reactive protein (CRP)
* Interferon-alpha, interleukin-6, interleukin-12, interferon-gamma, TNF-alpha (up-regulation of gene expression)
* Immunohistochemistry and characterization of cell types (CD8, T-cells, macrophages, dendritic cells)
* In addition, blood serum samples will be preserved and frozen for later tests that will be specified to the patients. The preserved material will be stored for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form.
* Male or non-pregnant, non-lactating female, ≥ 18 years.
* Must have a previously untreated, histologically confirmed nBCC on head, neck, trunk or arms.
* nBCC must not be larger than 20 mm in diameter and must be less than 5 mm in depth.
* Willing and able to participate in the trial as an outpatient and comply with all trial requirements.

Exclusion Criteria:

* nBCC located close to or at mouth or eyes.
* Patients who have had an organ transplant.
* Known autoimmune disorder (especially psoriasis), impaired immune system (e.g. HIV), known thyroid abnormalities, known depression.
* An open wound or an infection in treatment area.
* Dermatological disease or condition (e.g. rosacea, atopic dermatitis, eczema) in the treatment or surrounding area that might impair trial assessments.
* Evidence of an active infection or systemic cancer.
* Flu or flu-like symptoms (including general indisposition, fever, nausea, muscle pain, chills) within a week before start of the trial.
* Known allergy or hypersensitivity to any of the trial gel ingredients.
* Evidence of unstable or uncontrolled clinically significant medical conditions as determined by the investigator (e.g., renal or hepatic disease).
* Current alcohol abuse or chemical dependency as assessed by the investigator.
* Patient who is detained or committed to an institution by a law court or by legal authorities.
* Participation in another clinical trial within one month before start of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Dummer, PrMD, Principal Investigator — Clinical Dermatolgy Zurich
Locations (2):
- Hauttumorcentrum Charité (HTCC), Berlin, Germany
- Universitaetsspital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.06% Resiquimod Gel - A: * 60 mg gel
  * Once daily prior to normal sleeping hours
  * 5x within 1 week (Monday to Friday) for 4 weeks (at maximum) or until clinical manifestation of skin erosion/crust formation
  0.06% Resiquimod Gel - A
- 0.06% Resiquimod Gel - B: * 100 mg gel
  * Once daily prior to normal sleeping hours
  * 5x within 1 week (Monday to Friday) for 4 weeks (at maximum) or until clinical manifestation of skin erosion/crust formation
  0.06% Resiquimod Gel - B
- 0.06% Resiquimod Gel - C: * 100 mg gel
  * Once daily prior to normal sleeping hours
  * 5x within 1 week (Monday to Friday) for 4 weeks (at maximum) or until clinical manifestation of skin erosion/crust formation
  * The BCC will be pretreated. A shave biopsy (curettage or scraping off the tissue in a broad, superficial, tangential way) will be performed
  0.06% Resiquimod Gel - C
Period: Overall Study
Arm/Group | 0.06% Resiquimod Gel - A | 0.06% Resiquimod Gel - B | 0.06% Resiquimod Gel - C
Started | 1 | 3 | 0
Completed | 1 | 3 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.06% Resiquimod Gel - A | 0.06% Resiquimod Gel - B | 0.06% Resiquimod Gel - C | Total
Number analyzed (Participants) | 1 | 3 | 0 | 4
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 0 | 0 |  | 0
  >=65 years | 1 | 3 |  | 4
Gender [Number; unit: participants]
  Female | 0 | 1 |  | 1
  Male | 1 | 2 |  | 3
Region of Enrollment [Number; unit: participants]
  Switzerland | 1 | 3 |  | 4
  Germany | 0 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Histological Cure Rate
Time Frame: 8 weeks after a maximal treatment period of 4 weeks
Population: data were not collected for any of study participant.
Arm/Group | 0.06% Resiquimod Gel - A | 0.06% Resiquimod Gel - B | 0.06% Resiquimod Gel - C
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Complete Clinical Clearance Rate
Time Frame: 8 weeks after the 4 weeks treatment period
Population: data were not collected for any of study participant.
Groups:
- 0.06% Resiquimod Gel - C: * 100 mg gel
  * Once daily prior to normal sleeping hours
  * 5x within 1 week (Monday to Friday) for 4 weeks (at maximum) or until clinical manifestation of skin erosion/crust formation
  * The BCC will be pretreated. A shave biopsy (curettage or scraping off the tissue in a broad, superficial, tangential way) will be performed
  0.06% Resiquimod Gel - C: shave biopsy of BCC followed by single 100mg dose
Arm/Group | 0.06% Resiquimod Gel - A | 0.06% Resiquimod Gel - B | 0.06% Resiquimod Gel - C
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Evaluation of Local Tolerability by Means of 5-point Scales
Description: local skin reactions as erythema, edema, erosion/ulceration, exudate, dryness, encrustation judged by investigator by means of 5-point scales (0 = absent, 1 = slight, 2 = moderate, 3 = severe, 4 = very severe).
Time Frame: up to 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Evaluation of Systemic Tolerability Based on Haematology and Blood Chemistry Values and Vital Signs
Time Frame: up to 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Global Judgment of Tolerability by Investigator by Means of a 6-point Scale
Time Frame: 8 weeks after a maximal treatment period of 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 0.06% Resiquimod Gel - A | 0.06% Resiquimod Gel - B | 0.06% Resiquimod Gel - C
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 1/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.06% Resiquimod Gel - A (N=1) | 0.06% Resiquimod Gel - B (N=3) | 0.06% Resiquimod Gel - C (N=0)
Mutlilocular BCC right had Prox. (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nodular BCC arm left (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
superficial BCC submammary (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.06% Resiquimod Gel - A (N=1) | 0.06% Resiquimod Gel - B (N=3) | 0.06% Resiquimod Gel - C (N=0)
exertional dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
cornu cutaneum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator is granted a right to publish and present Trial Results together with other investigators of Trial and to be referred to in publications containing such results. However, investigator shall not publish or present Trial Results unless Investigator has submitted to Spirig a draft of the intended publication or presentation for review and approval.